CLINICAL TRIAL: NCT06608368
Title: A Randomized, Controlled Clinical Study Assessing the Effects of a Marketed Dentifrice Compared to a Regular Fluoride Dentifrice and a Positive Control Dentifrice on Tooth Sensitivity While Undergoing Tooth Bleaching
Brief Title: A Clinical Study Assessing the Effects of a Marketed Dentifrice on Tooth Sensitivity While Undergoing Tooth Bleaching
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300106
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Dentifrice (Experimental): Participants will dose the toothbrush provided with a strip of test dentifrice containing 5% weight by weight (w/w) NovaMin (Calcium Sodium Phosphosilicate) and 1040 parts per million (ppm) fluoride as sodium fluoride on each brushing occasion and will brush for one timed minute twice daily (morning and evening) for up to 5 weeks. Participants will use the dentifrice for 2 weeks pre tooth bleaching, 1 week during tooth bleaching and 2 weeks post tooth bleaching application. At Week 3, participants will perform the first application of tooth bleaching as per the instructions provided and continue the application once daily for up to 7 days.
  Interventions: Drug: Test Dentifrice (Sensodyne Repair and Protect Original Mint)
- Positive Control Dentifrice (Active Comparator): Participants will dose the toothbrush provided with a strip of positive control dentifrice containing 5% w/w KNO3 and 1150 ppm fluoride as sodium fluoride on each brushing occasion and will brush for one timed minute twice daily (morning and evening) for up to 5 weeks. Participants will use the dentifrice for 2 weeks pre tooth bleaching, 1 week during tooth bleaching and 2 weeks post tooth bleaching application. At Week 3, participants will perform the first application of tooth bleaching as per the instructions provided and continue the application once daily for up to 7 days.
  Interventions: Drug: Positive Control Dentifrice (Sensodyne Fresh Mint)
- Reference Dentifrice (Active Comparator): Participants will dose the toothbrush provided with a strip of reference dentifrice containing 1100 ppm fluoride as sodium fluoride on each brushing occasion and will brush for one timed minute twice daily (morning and evening) for up to 5 weeks. Participants will use the dentifrice for 2 weeks pre tooth bleaching, 1 week during tooth bleaching and 2 weeks post tooth bleaching application. At Week 3, participants will perform the first application of tooth bleaching as per the instructions provided and continue the application once daily for up to 7 days.
  Interventions: Drug: Reference Dentifrice (Crest Cavity Protection Regular)

INTERVENTIONS:
Drug: Test Dentifrice (Sensodyne Repair and Protect Original Mint) — Dentifrice containing 5% w/w NovaMin (Calcium Sodium Phosphosilicate) and 1040 ppm fluoride as sodium fluoride.
  Arms: Test Dentifrice
Drug: Positive Control Dentifrice (Sensodyne Fresh Mint) — Dentifrice containing 5% w/w KNO3 and 1150 ppm fluoride as sodium fluoride.
  Arms: Positive Control Dentifrice
Drug: Reference Dentifrice (Crest Cavity Protection Regular) — Dentifrice containing 1100 ppm fluoride as sodium fluoride.
  Arms: Reference Dentifrice

SUMMARY:
The aim of this study is to investigate the efficacy of a marketed dentifrice containing 5 percent (%) NovaMin (Calcium Sodium Phosphosilicate) to reduce tooth sensitivity during and post tooth bleaching compared to a marketed dentifrice containing 5% potassium nitrate (KNO3) and a marketed regular fluoride-containing dentifrice.

DETAILED DESCRIPTION:
This is a randomized, examiner blind, single-center, controlled, three arm, parallel group, proof-of-principal study to evaluate tooth sensitivity during and following a course of at-home tooth bleaching in participants with and without clinically confirmed dentine hypersensitivity (DH). The study will recruit generally healthy participants who wish to undergo peroxide tooth bleaching. Sufficient participants will be screened to randomize approximately 90 participants to study treatment (approximately 30 per treatment group).

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant is of either sex and any gender who, at the time of screening, is between the ages of 18-65 years, inclusive.
* Participant is willing and able to comply with scheduled visits, and other study procedures and restrictions.
* Participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history (for example, a medical condition confirmed to be causing xerostomia), or upon oral examination, that would impact the participant's safety, wellbeing or the outcomes of the study, if they were to participate in the study, or affect the participant's ability to understand and follow study procedures and requirements.
* Participant who wishes and is able to undergo at-home peroxide tooth bleaching.
* Participant with generally good oral health that fulfil all of the following:

  1. Having no lesions of the teeth or oral cavity that could interfere with the study evaluations.
  2. At least a total of 11 of the facial surfaces of maxillary and mandibular anterior 6 teeth (tooth numbers 6-11 and 22-27) suitable for peroxide whitening and gradable for VITA Bleachedguide evaluation with no significant defects, calculus, restorations, crowns or veneers that could impact tooth bleaching performance or study evaluations as judged by the clinical examiner.
  3. A minimum of 16 natural teeth.

Exclusion Criteria:

* Participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a Haleon employee directly involved in the conduct of the study or a member of their immediate family.
* Participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 60 days prior to study entry and/or during study participation.
* Participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* Participant who is pregnant or intending to become pregnant over the duration of the study or who is breastfeeding.
* Participant with known or suspected intolerance or hypersensitivity to the study materials [including the peroxide whitening gel] (or closely related compounds) or any of their stated ingredients.
* Participant who, in the opinion of the investigator or medically qualified designee, has a condition that would impact on their safety or wellbeing or affect their ability to understand and follow study procedures and requirements or who should not participate in the study for other reasons.
* Participant unwilling or unable to comply with the Lifestyle Considerations described in this protocol.
* Participant with a recent history (within the last year) of alcohol or other substance abuse.
* Participant with gross periodontal disease or who has had treatment for periodontal disease (including surgery) within 12 months of Screening or who has had scaling or root planning within 3 months of Screening.
* Participant who has had a tooth bleaching procedure (either professionally dispensed or at home) within 12 months of Screening.
* Participant with a fixed or removable partial prosthesis, multiple dental implants or orthodontic braces/bands or fixed retainer or togue/lip piercing which, in the opinion of the investigator, could impact study outcomes.
* During the period from screening till 2 weeks post completion of tooth bleaching, participant taking daily doses of medication/treatments which, in the opinion of the investigator or medically qualified designee, could interfere with their perception of tooth sensitivity (examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilizers, antidepressants, mood-altering and anti-inflammatory drugs).
* Participant who has previously been enrolled in this study.
* Participant who has used an oral care product indicated for the relief of DH or care of sensitive teeth within 8 weeks of Screening (participants will be required to verbally confirm the name of their current oral care products to enable site staff to verify the absence of known sensitivity ingredients).
* Participant who is taking daily doses of a medication which, in the opinion of the investigator or medically qualified designee, is causing xerostomia.
* Participant who has had dental prophylaxis within 4 weeks of Screening or who requires antibiotic prophylaxis for dental procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- All Sum Research, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in Canada.
Pre-assignment Details: A total of 91 participants were screened of which 90 participants were enrolled and randomized to receive treatment in 3 groups: Test Dentifrice (31 participants), Positive Control Dentifrice (29 participants), and Reference Dentifrice (30 participants). A total of 88 participants completed the study.
Groups:
- Test Dentifrice (NovaMin Containing Dentifrice): Participants dosed the toothbrush provided with a strip of Test dentifrice containing 5 percent (%) weight by weight (w/w) NovaMin (Calcium Sodium Phosphosilicate) and 1040 parts per million (ppm) fluoride as sodium fluoride on each brushing occasion and brushed their teeth for one timed minute twice daily (morning and evening) for up to 5 weeks. Participants used the dentifrice for 2 weeks pre tooth bleaching, 1 week during tooth bleaching and 2 weeks post tooth bleaching application. At Week 3, participants performed the first application of tooth bleaching as per the instructions provided and continued the application once daily for up to 7 days.
- Positive Control Dentifrice (KNO3 Containing Dentifrice): Participants dosed the toothbrush provided with a strip of Positive Control dentifrice containing 5% w/w KNO3 and 1150 ppm fluoride as sodium fluoride on each brushing occasion and brushed their teeth for one timed minute twice daily (morning and evening) for up to 5 weeks. Participants used the dentifrice for 2 weeks pre tooth bleaching, 1 week during tooth bleaching and 2 weeks post tooth bleaching application. At Week 3, participants performed the first application of tooth bleaching as per the instructions provided and continued the application once daily for up to 7 days.
- Reference Dentifrice (Regular Fluoride Dentifrice): Participants dosed the toothbrush provided with a strip of Reference dentifrice containing 1100 ppm fluoride as sodium fluoride on each brushing occasion and brushed their teeth for one timed minute twice daily (morning and evening) for up to 5 weeks. Participants used the dentifrice for 2 weeks pre tooth bleaching, 1 week during tooth bleaching and 2 weeks post tooth bleaching application. At Week 3, participants performed the first application of tooth bleaching as per the instructions provided and continued the application once daily for up to 7 days.
Period: Overall Study
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Started | 31 | 29 | 30
Completed | 31 | 27 | 30
Not Completed | 0 | 2 | 0
Not completed — Family Emergency | 0 | 1 | 0
Not completed — Scheduling Issues | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least one dose of the study product.
Groups:
- Test Dentifrice (NovaMin Containing Dentifrice): Participants dosed the toothbrush provided with a strip of Test dentifrice containing 5% w/w NovaMin (Calcium Sodium Phosphosilicate) and 1040 ppm fluoride as sodium fluoride on each brushing occasion and brushed their teeth for one timed minute twice daily (morning and evening) for up to 5 weeks. Participants used the dentifrice for 2 weeks pre tooth bleaching, 1 week during tooth bleaching and 2 weeks post tooth bleaching application. At Week 3, participants performed the first application of tooth bleaching as per the instructions provided and continued the application once daily for up to 7 days.
- Total: Total of all reporting groups
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice) | Total
Number analyzed (Participants) | 31 | 29 | 30 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (14.46) | 48.8 (13.02) | 50.3 (9.25) | 48.3 (12.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 20 | 64
  Male | 10 | 6 | 10 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 3 | 3
  Not Hispanic or Latino | 31 | 29 | 27 | 87
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian and Alaskan Native | 1 | 0 | 0 | 1
  Asian | 3 | 2 | 7 | 12
  Black/African American | 12 | 11 | 14 | 37
  Other | 0 | 0 | 1 | 1
  White | 15 | 16 | 8 | 39

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS) Scores of the Tooth Sensitivity Questionnaire Collected Through the Study
Description: The tooth sensitivity questionnaire including the VAS was used to describe the overall tooth sensitivity experienced by the participant. Participants indicated whether they felt tooth sensitivity during the previous 24 hours using a Yes/No response. Participants who indicated they felt tooth sensitivity completed the remainder of the questionnaire and rated their overall tooth sensitivity using a 100 millimeter (mm) VAS with scores ranging from 0 mm (No Sensitivity) to 100 mm (Extreme Sensitivity). Participants made a single vertical mark at the point on the scale which represented the degree of overall tooth sensitivity (example twinges, pain and other sensations in their teeth) that they experienced over the last 24 hours. The marked-off line segment was measured in 'mm'. Lower scores indicated an improvement in sensitivity.
Time Frame: Up to Day 36
Population: Modified Intent-To-Treat (mITT) population included all randomized participants who completed at least one use of study product and had at least one VAS score for tooth sensitivity recorded during the tooth-bleaching period. Only those participants with data available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Number analyzed (Participants) | 31 | 27 | 30
millimeter
  Screening | 33.8 (37.00) | 41.6 (38.71) | 36.9 (38.73)
  Baseline | 31.1 (35.07) | 36.9 (36.09) | 36.5 (38.54)
  Bleaching Period: Day 1: number analyzed (Participants) | 26 | 22 | 24
  Bleaching Period: Day 1 | 34.3 (34.24) | 34.9 (35.35) | 37.1 (38.72)
  Bleaching Period: Day 2 | 38.0 (36.65) | 35.9 (36.41) | 36.2 (35.88)
  Bleaching Period: Day 3 | 37.5 (35.54) | 33.9 (36.08) | 35.3 (32.54)
  Bleaching Period: Day 4 | 39.7 (36.03) | 36.1 (34.51) | 39.7 (34.44)
  Bleaching Period: Day 5 | 33.3 (35.66) | 38.6 (34.52) | 34.9 (35.00)
  Bleaching Period: Day 6 | 34.0 (33.89) | 37.7 (35.04) | 33.9 (34.95)
  Bleaching Period: Day 7 | 34.0 (34.91) | 37.1 (34.79) | 31.9 (35.32)
  Post Bleaching Period: Day 1 | 28.3 (31.48) | 30.1 (32.43) | 30.2 (35.82)
  Post Bleaching Period: Day 2 | 27.2 (32.33) | 26.9 (31.65) | 29.9 (35.77)
  Post Bleaching Period: Day 3 | 23.8 (30.72) | 23.6 (30.15) | 29.5 (35.28)
  Post Bleaching Period: Day 4 | 24.9 (31.16) | 23.8 (30.21) | 28.4 (33.89)
  Post Bleaching Period: Day 5 | 22.5 (30.48) | 22.4 (29.48) | 28.4 (33.64)
  Post Bleaching Period: Day 6 | 22.7 (30.66) | 23.1 (29.74) | 28.3 (33.58)
  Post Bleaching Period: Day 7 | 22.1 (30.16) | 21.3 (29.32) | 28.0 (33.52)
  Post Bleaching Period: Day 8 | 21.0 (28.58) | 21.8 (30.41) | 27.7 (33.41)
  Post Bleaching Period: Day 9 | 22.3 (29.77) | 18.9 (28.57) | 27.9 (33.47)
  Post Bleaching Period: Day 10 | 22.4 (29.81) | 17.7 (27.96) | 26.7 (32.75)
  Post Bleaching Period: Day 11 | 20.9 (29.40) | 18.1 (28.59) | 26.9 (32.39)
  Post Bleaching Period: Day 12 | 19.9 (29.09) | 17.6 (28.26) | 27.6 (33.18)
  Post Bleaching Period: Day 13 | 19.3 (28.12) | 17.3 (28.21) | 27.8 (33.68)
  Post Bleaching Period: Day 14 | 20.1 (28.38) | 18.3 (28.72) | 26.9 (32.52)

2. Primary Outcome: Labelled Magnitude Scale (LMS) Scores of the Tooth Sensitivity Questionnaire Collected Through the Study: Intensity
Description: The tooth sensitivity questionnaire including the LMS was used to describe the overall tooth sensitivity experienced by the participants. Participants indicated whether they felt tooth sensitivity during the previous 24 hours using a Yes/No response. Participants with a Yes response completed the remainder of the questionnaire and rated the intensity of their tooth sensitivity using the individual 100 mm LMS for intensity. The scale was labelled with descriptive words related to intensity and ranged from 0 mm to 100 mm where lower scores indicated better outcome (no pain). Participants marked the scale to indicate the best description of the intensity of their sensitivity and the marked-off line segment was measured in 'mm'. Lower scores indicated an improvement in sensitivity.
Time Frame: Up to Day 36
Population: mITT population. Only those participants with data available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Number analyzed (Participants) | 31 | 27 | 30
millimeter
  Screening | 28.1 (30.95) | 38.8 (35.79) | 32.6 (35.57)
  Baseline | 26.5 (29.76) | 34.1 (33.49) | 33.0 (36.02)
  Bleaching Period: Day 1: number analyzed (Participants) | 26 | 22 | 24
  Bleaching Period: Day 1 | 29.7 (29.82) | 33.3 (34.07) | 31.6 (35.60)
  Bleaching Period: Day 2 | 30.5 (30.83) | 30.1 (31.85) | 33.4 (33.14)
  Bleaching Period: Day 3 | 30.0 (29.04) | 29.4 (31.34) | 33.3 (29.92)
  Bleaching Period: Day 4 | 30.4 (29.13) | 30.9 (28.96) | 35.5 (30.36)
  Bleaching Period: Day 5 | 25.9 (28.92) | 31.7 (28.86) | 29.2 (28.48)
  Bleaching Period: Day 6 | 26.2 (26.59) | 30.0 (27.68) | 26.6 (27.06)
  Bleaching Period: Day 7 | 26.1 (27.19) | 28.5 (28.68) | 26.0 (28.62)
  Post Bleaching Period: Day 1 | 21.6 (24.47) | 25.4 (28.80) | 23.7 (28.05)
  Post Bleaching Period: Day 2 | 20.8 (23.97) | 23.7 (28.36) | 23.1 (28.21)
  Post Bleaching Period: Day 3 | 19.8 (23.83) | 22.4 (26.93) | 23.5 (27.19)
  Post Bleaching Period: Day 4 | 17.5 (21.53) | 21.3 (27.02) | 22.0 (27.43)
  Post Bleaching Period: Day 5 | 16.5 (21.01) | 20.7 (27.01) | 21.3 (25.67)
  Post Bleaching Period: Day 6 | 17.1 (21.16) | 20.8 (25.79) | 20.3 (25.72)
  Post Bleaching Period: Day 7 | 16.2 (20.66) | 19.2 (25.11) | 19.4 (25.85)
  Post Bleaching Period: Day 8 | 15.5 (20.59) | 18.7 (25.58) | 20.2 (25.96)
  Post Bleaching Period: Day 9 | 15.4 (20.53) | 16.9 (24.29) | 19.7 (25.99)
  Post Bleaching Period: Day 10 | 15.1 (20.52) | 16.6 (24.32) | 19.3 (25.84)
  Post Bleaching Period: Day 11 | 15.3 (20.68) | 16.0 (24.50) | 18.7 (25.22)
  Post Bleaching Period: Day 12 | 14.9 (20.30) | 15.2 (23.62) | 18.2 (25.13)
  Post Bleaching Period: Day 13 | 15.1 (19.76) | 14.4 (23.18) | 18.5 (25.35)
  Post Bleaching Period: Day 14 | 15.2 (20.10) | 14.9 (23.81) | 18.6 (25.38)

3. Primary Outcome: LMS Scores of the Tooth Sensitivity Questionnaire Collected Through the Study: Duration
Description: The tooth sensitivity questionnaire including the LMS was used to describe the overall tooth sensitivity experienced by the participants. Participants indicated whether they felt tooth sensitivity during the previous 24 hours using a Yes/No response. Participants with a Yes response completed the remainder of the questionnaire and rated the duration of their tooth sensitivity using the individual 100 mm LMS for duration. The scale was labelled with descriptive words related to duration and ranged from 0 mm to 100 mm where lower scores indicated better outcome (no pain). Participants marked the scale to indicate the best description of the duration of sensitivity and the marked-off line segment was measured in 'mm'. Lower scores indicated an improvement in sensitivity.
Time Frame: Up to Day 36
Population: mITT population. Only those participants with data available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Number analyzed (Participants) | 31 | 27 | 30
millimeter
  Screening | 18.8 (21.55) | 26.4 (25.30) | 24.4 (26.28)
  Baseline | 18.0 (21.55) | 23.0 (22.19) | 24.6 (26.76)
  Bleaching Period: Day 1: number analyzed (Participants) | 26 | 22 | 24
  Bleaching Period: Day 1 | 19.7 (22.14) | 21.7 (21.33) | 23.6 (25.56)
  Bleaching Period: Day 2 | 23.5 (24.45) | 20.7 (21.66) | 26.6 (25.74)
  Bleaching Period: Day 3 | 23.2 (22.58) | 22.4 (23.66) | 31.2 (25.29)
  Bleaching Period: Day 4 | 23.9 (22.94) | 26.0 (22.18) | 29.7 (25.00)
  Bleaching Period: Day 5 | 20.0 (21.96) | 26.7 (23.24) | 27.0 (25.43)
  Bleaching Period: Day 6 | 23.5 (21.55) | 28.7 (24.22) | 25.9 (24.33)
  Bleaching Period: Day 7 | 21.7 (21.87) | 28.2 (25.51) | 24.5 (24.89)
  Post Bleaching Period: Day 1 | 18.5 (20.71) | 24.5 (24.16) | 23.8 (25.35)
  Post Bleaching Period: Day 2 | 16.8 (20.80) | 22.2 (23.45) | 22.3 (24.65)
  Post Bleaching Period: Day 3 | 17.1 (21.53) | 20.7 (21.64) | 23.5 (24.80)
  Post Bleaching Period: Day 4 | 15.1 (20.13) | 18.9 (20.89) | 22.4 (24.71)
  Post Bleaching Period: Day 5 | 15.8 (21.35) | 17.7 (20.60) | 22.4 (24.41)
  Post Bleaching Period: Day 6 | 15.4 (20.35) | 18.9 (21.52) | 20.5 (24.08)
  Post Bleaching Period: Day 7 | 15.1 (20.42) | 18.4 (21.48) | 19.1 (23.14)
  Post Bleaching Period: Day 8 | 14.8 (20.17) | 16.9 (19.92) | 18.4 (22.51)
  Post Bleaching Period: Day 9 | 13.9 (19.28) | 13.9 (19.30) | 18.3 (22.41)
  Post Bleaching Period: Day 10 | 14.4 (19.85) | 13.6 (19.38) | 17.7 (22.47)
  Post Bleaching Period: Day 11 | 14.6 (20.08) | 13.7 (19.92) | 17.6 (22.05)
  Post Bleaching Period: Day 12 | 14.1 (19.71) | 13.1 (19.29) | 17.5 (22.53)
  Post Bleaching Period: Day 13 | 13.9 (19.34) | 13.0 (19.08) | 17.5 (22.04)
  Post Bleaching Period: Day 14 | 15.2 (20.07) | 13.4 (18.70) | 17.4 (21.80)

4. Primary Outcome: LMS Scores of the Tooth Sensitivity Questionnaire Collected Through the Study: Tolerability
Description: The tooth sensitivity questionnaire including the LMS was used to describe the overall tooth sensitivity experienced by the participants. Participants indicated whether they felt tooth sensitivity during the previous 24 hours using a Yes/No response. Participants with a 'Yes' response completed the remainder of the questionnaire and rated the tolerability of their tooth sensitivity using the individual 100 mm LMS for tolerability. The scale was labelled with descriptive words related to tolerability and ranged from 0 mm to 100 mm where lower scores indicated better outcome (no pain). Participants marked the scale to indicate the best description of the tolerability of their sensitivity and the marked-off line segment was measured in 'mm'. Lower scores indicated an improvement in sensitivity.
Time Frame: Upto Day 36
Population: mITT population. Only those participants with data available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Number analyzed (Participants) | 31 | 27 | 30
millimeter
  Screening | 20.7 (25.13) | 21.9 (22.88) | 19.9 (22.37)
  Baseline | 19.4 (24.84) | 20.9 (22.56) | 21.0 (23.95)
  Baseline Period: Day 1: number analyzed (Participants) | 26 | 22 | 24
  Baseline Period: Day 1 | 22.6 (24.42) | 19.9 (22.93) | 22.2 (24.50)
  Baseline Period: Day 2 | 24.1 (27.44) | 19.8 (22.66) | 22.3 (23.68)
  Baseline Period: Day 3 | 23.8 (25.83) | 21.9 (24.65) | 22.8 (21.55)
  Baseline Period: Day 4 | 23.7 (25.87) | 22.8 (22.54) | 25.0 (22.96)
  Baseline Period: Day 5 | 21.5 (25.25) | 23.6 (22.85) | 22.9 (23.81)
  Baseline Period: Day 6 | 23.4 (24.18) | 24.1 (24.53) | 22.4 (23.49)
  Baseline Period: Day 7 | 22.6 (24.72) | 24.6 (26.02) | 21.5 (24.76)
  Post Baseline Period: Day 1 | 18.0 (21.53) | 20.5 (25.84) | 20.5 (25.43)
  Post Baseline Period: Day 2 | 17.0 (21.21) | 20.7 (26.21) | 19.3 (24.72)
  Post Baseline Period: Day 3 | 15.5 (20.91) | 19.4 (25.28) | 21.7 (25.21)
  Post Baseline Period: Day 4 | 15.5 (20.71) | 18.3 (24.70) | 19.6 (24.34)
  Post Baseline Period: Day 5 | 14.4 (19.76) | 16.8 (24.32) | 18.6 (23.80)
  Post Baseline Period: Day 6 | 14.7 (19.94) | 17.9 (24.36) | 19.1 (24.64)
  Post Baseline Period: Day 7 | 14.2 (19.91) | 15.4 (22.57) | 17.5 (23.71)
  Post Baseline Period: Day 8 | 14.5 (20.21) | 17.9 (23.64) | 17.5 (23.27)
  Post Baseline Period: Day 9 | 14.7 (20.41) | 13.8 (20.75) | 17.0 (23.13)
  Post Baseline Period: Day 10 | 14.4 (19.86) | 13.3 (20.37) | 15.9 (22.53)
  Post Baseline Period: Day 11 | 13.9 (20.20) | 12.6 (20.29) | 16.1 (22.58)
  Post Baseline Period: Day 12 | 13.8 (19.94) | 11.7 (19.02) | 15.9 (22.73)
  Post Baseline Period: Day 13 | 13.5 (19.82) | 11.9 (19.31) | 16.2 (22.77)
  Post Baseline Period: Day 14 | 14.2 (20.11) | 12.4 (20.07) | 16.0 (22.67)

5. Primary Outcome: LMS Scores of the Tooth Sensitivity Questionnaire Collected Through the Study: Description
Description: The tooth sensitivity questionnaire including the LMS was used to describe the overall tooth sensitivity experienced by the participants. Participants indicated whether they felt tooth sensitivity during the previous 24 hours using a Yes/No response. Participants with a 'Yes' response completed the remainder of the questionnaire and rated the tolerability of their tooth sensitivity using the individual 100 mm LMS for description. The scale was labelled with descriptive words related to the quality of tooth sensitivity and ranged from 0 mm to 100 mm where lower scores indicated better outcome (no pain). Participants marked the scale to indicate the best description of their sensitivity and the marked-off line segment was measured in 'mm'. Lower scores indicated an improvement in sensitivity.
Time Frame: Up to Day 36
Population: mITT Population. Only those participants with data available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Number analyzed (Participants) | 31 | 27 | 30
millimeter
  Screening | 28.8 (35.71) | 36.4 (38.09) | 35.2 (38.67)
  Baseline | 27.4 (34.75) | 32.2 (35.28) | 34.6 (38.33)
  Baseline Period: Day 1: number analyzed (Participants) | 26 | 22 | 24
  Baseline Period: Day 1 | 29.3 (34.81) | 30.5 (35.70) | 33.3 (38.06)
  Baseline Period: Day 2 | 31.0 (34.60) | 28.2 (33.82) | 33.0 (34.47)
  Baseline Period: Day 3 | 33.4 (36.27) | 27.9 (31.99) | 37.0 (32.25)
  Baseline Period: Day 4 | 31.3 (33.33) | 33.3 (30.62) | 40.7 (34.32)
  Baseline Period: Day 5 | 28.7 (33.43) | 31.0 (29.59) | 31.8 (32.17)
  Baseline Period: Day 6 | 29.2 (31.35) | 31.8 (28.97) | 30.9 (30.74)
  Baseline Period: Day 7 | 28.2 (31.93) | 30.1 (28.26) | 28.3 (31.04)
  Post Baseline Period: Day 1 | 23.6 (28.71) | 28.4 (30.35) | 24.6 (29.32)
  Post Baseline Period: Day 2 | 22.1 (28.49) | 26.6 (28.98) | 23.9 (29.11)
  Post Baseline Period: Day 3 | 20.8 (27.25) | 25.5 (28.77) | 25.6 (28.87)
  Post Baseline Period: Day 4 | 19.3 (26.64) | 24.2 (28.34) | 24.0 (28.75)
  Post Baseline Period: Day 5 | 18.6 (25.52) | 21.9 (27.04) | 23.9 (28.53)
  Post Baseline Period: Day 6 | 19.9 (25.90) | 21.7 (25.24) | 21.2 (27.08)
  Post Baseline Period: Day 7 | 18.2 (25.32) | 19.2 (23.23) | 21.3 (27.70)
  Post Baseline Period: Day 8 | 17.6 (25.19) | 19.8 (24.09) | 21.4 (27.90)
  Post Baseline Period: Day 9 | 17.8 (25.64) | 16.1 (21.47) | 21.4 (28.09)
  Post Baseline Period: Day 10 | 17.4 (24.66) | 16.7 (22.20) | 20.5 (27.74)
  Post Baseline Period: Day 11 | 17.2 (24.85) | 14.7 (21.38) | 20.6 (28.00)
  Post Baseline Period: Day 12 | 17.2 (24.72) | 15.4 (23.36) | 19.5 (26.89)
  Post Baseline Period: Day 13 | 17.5 (24.01) | 14.0 (20.98) | 19.9 (27.16)
  Post Baseline Period: Day 14 | 17.6 (24.05) | 14.5 (20.97) | 19.6 (27.00)

6. Primary Outcome: Bothersomeness Numerical Rating Scale (NRS) Score of Tooth Sensitivity Questionnaire Collected Through the Study
Description: The tooth sensitivity questionnaire including Bothersomeness NRS was used to describe the overall tooth sensitivity experienced by the participant. Participants indicated whether they felt tooth sensitivity during the previous 24 hours. Participants who indicated they felt tooth sensitivity completed the remainder of the questionnaire and rated how bothered they had been by any tooth sensitivity (example twinges, pain, ache or other sensations in teeth) using the Bothersomeness NRS scale. The scale ranged from 1 (Not bothered at all) to 10 (Extremely bothered). Lower scores indicated an improvement in sensitivity.
Time Frame: Up to Day 36
Population: mITT population. Only those participants with data available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Number analyzed (Participants) | 31 | 27 | 30
score on a scale
  Screening | 3.5 (2.85) | 3.9 (2.86) | 4.1 (3.28)
  Baseline | 3.2 (2.56) | 3.4 (2.60) | 4.1 (3.30)
  Baseline Period: Day 1: number analyzed (Participants) | 26 | 22 | 24
  Baseline Period: Day 1 | 3.5 (2.70) | 3.3 (2.66) | 4.1 (3.23)
  Baseline Period: Day 2 | 3.7 (2.81) | 3.3 (2.57) | 4.3 (3.27)
  Baseline Period: Day 3 | 3.9 (2.79) | 3.3 (2.70) | 4.3 (3.03)
  Baseline Period: Day 4 | 3.9 (2.79) | 3.3 (2.48) | 4.5 (3.07)
  Baseline Period: Day 5 | 3.5 (2.78) | 3.5 (2.62) | 4.2 (3.15)
  Baseline Period: Day 6 | 3.7 (2.67) | 3.5 (2.75) | 4.0 (3.13)
  Baseline Period: Day 7 | 3.5 (2.67) | 3.6 (2.74) | 3.9 (3.13)
  Post Baseline Period: Day 1 | 3.3 (2.49) | 3.2 (2.59) | 3.6 (3.11)
  Post Baseline Period: Day 2 | 3.1 (2.46) | 3.1 (2.58) | 3.6 (3.12)
  Post Baseline Period: Day 3 | 2.9 (2.39) | 3.0 (2.53) | 3.7 (3.11)
  Post Baseline Period: Day 4 | 2.9 (2.37) | 2.9 (2.56) | 3.5 (2.97)
  Post Baseline Period: Day 5 | 2.7 (2.31) | 2.9 (2.41) | 3.5 (2.98)
  Post Baseline Period: Day 6 | 2.7 (2.29) | 2.9 (2.41) | 3.4 (2.95)
  Post Baseline Period: Day 7 | 2.6 (2.29) | 2.7 (2.40) | 3.4 (2.97)
  Post Baseline Period: Day 8 | 2.7 (2.26) | 2.8 (2.41) | 3.4 (2.92)
  Post Baseline Period: Day 9 | 2.7 (2.27) | 2.5 (2.21) | 3.4 (2.88)
  Post Baseline Period: Day 10 | 2.6 (2.17) | 2.5 (2.17) | 3.3 (2.87)
  Post Baseline Period: Day 11 | 2.6 (2.17) | 2.5 (2.24) | 3.3 (2.84)
  Post Baseline Period: Day 12 | 2.5 (2.22) | 2.5 (2.21) | 3.3 (2.88)
  Post Baseline Period: Day 13 | 2.5 (2.19) | 2.4 (2.22) | 3.3 (2.81)
  Post Baseline Period: Day 14 | 2.6 (2.16) | 2.5 (2.24) | 3.2 (2.75)

7. Primary Outcome: Number of Participants With a Tooth Sensitivity-free Day Through the Study
Description: Participants indicated whether they felt tooth sensitivity during the previous 24 hours as a Yes/No response in the tooth sensitivity questionnaire. Number of participants with 'No' response were reported.
Time Frame: Up to Day 36
Population: mITT population. Only those participants with data available at the specified time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Number analyzed (Participants) | 31 | 27 | 30
Participants
  Screening | 16 | 12 | 15
  Baseline | 16 | 12 | 15
  Bleaching Period: Day 1: number analyzed (Participants) | 26 | 22 | 24
  Bleaching Period: Day 1 | 12 | 10 | 12
  Bleaching Period: Day 2 | 14 | 13 | 13
  Bleaching Period: Day 3 | 12 | 13 | 10
  Bleaching Period: Day 4 | 12 | 9 | 10
  Bleaching Period: Day 5 | 12 | 9 | 12
  Bleaching Period: Day 6 | 10 | 8 | 11
  Bleaching Period: Day 7 | 11 | 8 | 13
  Post Bleaching Period: Day 1 | 12 | 10 | 14
  Post Bleaching Period: Day 2 | 14 | 11 | 14
  Post Bleaching Period: Day 3 | 16 | 11 | 14
  Post Bleaching Period: Day 4 | 15 | 12 | 15
  Post Bleaching Period: Day 5 | 17 | 12 | 15
  Post Bleaching Period: Day 6 | 16 | 11 | 16
  Post Bleaching Period: Day 7 | 16 | 11 | 15
  Post Bleaching Period: Day 8 | 17 | 11 | 16
  Post Bleaching Period: Day 9 | 16 | 14 | 16
  Post Bleaching Period: Day 10 | 16 | 14 | 17
  Post Bleaching Period: Day 11 | 17 | 15 | 16
  Post Bleaching Period: Day 12 | 17 | 15 | 17
  Post Bleaching Period: Day 13 | 16 | 15 | 17
  Post Bleaching Period: Day 14 | 16 | 14 | 17

8. Primary Outcome: Number of Participants Who Use Analgesics to Alleviate Tooth Sensitivity
Description: Participants indicated whether they used any pain killing medications to relieve tooth sensitivity/pain in the last 24 hours as a Yes/No response in the tooth sensitivity questionnaire. Number of participants with 'Yes' response were to be reported.
Time Frame: Up to Day 36
Population: mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Number analyzed (Participants) | 31 | 27 | 30
Participants | 0 | 0 | 0

9. Secondary Outcome: Mean VAS Score During Tooth Bleaching
Description: The tooth sensitivity questionnaire including the VAS was used to describe the overall tooth sensitivity experienced by the participant. Participants indicated whether they felt tooth sensitivity during the previous 24 hours using a Yes/No response. Participants who indicated that they felt tooth sensitivity completed the remainder of the questionnaire and rated their overall tooth sensitivity using a 100 mm VAS with scores ranging from 0 mm (No Sensitivity) to 100 mm (Extreme Sensitivity). Participants made a single vertical mark at the point on the scale which represented the degree of overall tooth sensitivity (example twinges, pain and other sensations in their teeth) that they experienced over the last 24 hours. The marked-off line segment was measured in 'mm'. Lower scores indicated an improvement in sensitivity.
Time Frame: Day 15 up to Day 21
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: millimeter
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Number analyzed (Participants) | 31 | 27 | 30
millimeter | 39.0423 (2.7961) | 32.8316 (2.9787) | 35.7939 (2.8196)
Statistical Analysis 1: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Positive Control Dentifrice (KNO3 Containing Dentifrice); Test type: Superiority; p = 0.1332, Mixed Model with Repeated Measures; Least Square Mean Difference = -6.2108, 95% CI 2-sided [-14.3568 to 1.9353], Standard Error of Mean 4.0959 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Test Dentifrice value
Statistical Analysis 2: Comparison: Positive Control Dentifrice (KNO3 Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); Test type: Superiority; p = 0.4722, Mixed Model with Repeated Measures; Least Square Mean Difference = -2.9623, 95% CI 2-sided [-11.1207 to 5.1960], Standard Error of Mean 4.1021 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Reference Dentifrice value
Statistical Analysis 3: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); Test type: Superiority; p = 0.4155, Mixed Model with Repeated Measures; Least Square Mean Difference = 3.2484, 95% CI 2-sided [-4.6456 to 11.1425], Standard Error of Mean 3.9692 — Least Square Mean Difference was calculated as Test Dentifrice value minus Reference Dentifrice value

10. Secondary Outcome: Mean LMS Score During Tooth Bleaching
Description: The tooth sensitivity questionnaire including the LMS was used to describe the overall tooth sensitivity experienced by the participant. Participants indicated whether they felt tooth sensitivity during the previous 24 hours using a Yes/No response. Participants who indicated they felt tooth sensitivity completed the remainder of the questionnaire and rated the intensity, duration, tolerability and descriptive quality of their tooth sensitivity using the four individual 100 mm LMS. Each individual scale was labelled with descriptive words related to the intensity, duration, tolerability, quality of tooth sensitivity and ranged from 0 mm to 100 mm where lower scores indicated better outcome (no pain). Participants marked each scale to indicate the best description of their sensitivity and the marked-off line segment was measured in 'mm'. Lower scores indicated an improvement in sensitivity.
Time Frame: Day 15 up to Day 21
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: millimeter
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Number analyzed (Participants) | 31 | 27 | 30
millimeter
  LMS Intensity | 31.4069 (2.2894) | 26.6679 (2.4227) | 31.1071 (2.2738)
  LMS Duration | 25.2392 (2.2168) | 22.5202 (2.3259) | 26.2188 (2.2087)
  LMS Tolerability | 23.3203 (2.0242) | 21.4742 (2.1743) | 23.5177 (2.0578)
  LMS Description | 33.2256 (2.7497) | 28.3419 (2.9352) | 32.3172 (2.7867)
Statistical Analysis 1: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Positive Control Dentifrice (KNO3 Containing Dentifrice); LMS Intensity; Test type: Superiority; p = 0.1650, Mixed Model with Repeated Measures; Least Square Mean Difference = -4.7390, 95% CI 2-sided [-11.4672 to 1.9891], Standard Error of Mean 3.3830 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Test Dentifrice value
Statistical Analysis 2: Comparison: Positive Control Dentifrice (KNO3 Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); LMS Intensity; Test type: Superiority; p = 0.1855, Mixed Model with Repeated Measures; Least Square Mean Difference = -4.4392, 95% CI 2-sided [-11.0516 to 2.1732], Standard Error of Mean 3.3248 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Reference Dentifrice value
Statistical Analysis 3: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); LMS Intensity; Test type: Superiority; p = 0.9261, Mixed Model with Repeated Measures; Least Square Mean Difference = 0.2998, 95% CI 2-sided [-6.1107 to 6.7104], Standard Error of Mean 3.2234 — Least Square Mean Difference was calculated as Test Dentifrice value minus Reference Dentifrice value
Statistical Analysis 4: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Positive Control Dentifrice (KNO3 Containing Dentifrice); LMS Duration; Test type: Superiority; p = 0.4039, Mixed Model with Repeated Measures; Least Square Mean Difference = -2.7189, 95% CI 2-sided [-9.1643 to 3.7265], Standard Error of Mean 3.2406 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Test Dentifrice value
Statistical Analysis 5: Comparison: Positive Control Dentifrice (KNO3 Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); LMS Duration; Test type: Superiority; p = 0.2505, Mixed Model with Repeated Measures; Least Square Mean Difference = -3.6986, 95% CI 2-sided [-10.0548 to 2.6577], Standard Error of Mean 3.1959 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Reference Dentifrice value
Statistical Analysis 6: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); LMS Duration; Test type: Superiority; p = 0.7577, Mixed Model with Repeated Measures; Least Square Mean Difference = -0.9797, 95% CI 2-sided [-7.2744 to 5.3151], Standard Error of Mean 3.1648 — Least Square Mean Difference was calculated as Test Dentifrice value minus Reference Dentifrice value
Statistical Analysis 7: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Positive Control Dentifrice (KNO3 Containing Dentifrice); LMS Tolerability; Test type: Superiority; p = 0.5367, Mixed Model with Repeated Measures; Least Square Mean Difference = -1.8461, 95% CI 2-sided [-7.7642 to 4.0720], Standard Error of Mean 2.9755 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Test Dentifrice value
Statistical Analysis 8: Comparison: Positive Control Dentifrice (KNO3 Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); LMS Tolerability; Test type: Superiority; p = 0.4963, Mixed Model with Repeated Measures; Least Square Mean Difference = -2.0435, 95% CI 2-sided [-7.9916 to 3.9047], Standard Error of Mean 2.9907 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Reference Dentifrice value
Statistical Analysis 9: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); LMS Tolerability; Test type: Superiority; p = 0.9457, Mixed Model with Repeated Measures; Least Square Mean Difference = -0.1974, 95% CI 2-sided [-5.9429 to 5.5481], Standard Error of Mean 2.8888 — Mean Difference was calculated as Test Dentifrice value minus Reference Dentifrice value
Statistical Analysis 10: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Positive Control Dentifrice (KNO3 Containing Dentifrice); LMS Description; Test type: Superiority; p = 0.2281, Mixed Model with Repeated Measures; Least Square Mean Difference = -4.8837, 95% CI 2-sided [-12.8837 to 3.1163], Standard Error of Mean 4.0222 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Test Dentifrice value
Statistical Analysis 11: Comparison: Positive Control Dentifrice (KNO3 Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); LMS Description; Test type: Superiority; p = 0.3290, Mixed Model with Repeated Measures; Least Square Mean Difference = -3.9754, 95% CI 2-sided [-12.0283 to 4.0775], Standard Error of Mean 4.0489 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Reference Dentifrice value
Statistical Analysis 12: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); LMS Description; Test type: Superiority; p = 0.8178, Mixed Model with Repeated Measures; Least Square Mean Difference = 0.9083, 95% CI 2-sided [-6.9076 to 8.7243], Standard Error of Mean 3.9297 — Least Square Mean Difference was calculated as Test Dentifrice value minus Reference Dentifrice value

11. Secondary Outcome: Mean Bothersomeness NRS Score During Tooth Bleaching
Description: The tooth sensitivity questionnaire was used to describe the overall tooth sensitivity experienced by the participant. Participants indicated whether they felt tooth sensitivity during the previous 24 hours. Participants who indicated they felt tooth sensitivity completed the remainder of the questionnaire and rated how bothered they were by any tooth sensitivity (example twinges, pain, ache or other sensations in teeth) using the Bothersomeness NRS scale. The scale ranged from 1 (Not bothered at all) to 10 (Extremely bothered). Lower scores indicated an improvement in sensitivity.
Time Frame: Day 15 up to Day 21
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Number analyzed (Participants) | 31 | 27 | 30
score on a scale | 3.9603 (0.2408) | 3.3288 (0.2581) | 3.9735 (0.2456)
Statistical Analysis 1: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Positive Control Dentifrice (KNO3 Containing Dentifrice); Test type: Superiority; p = 0.0756, Mixed Model with Repeated Measures; Least Square Mean Difference = -0.6315, 95% CI 2-sided [-1.3296 to 0.06658], Standard Error of Mean 0.3510 — Mean Difference was calculated as Positive Control Dentifrice value minus Test Dentifrice value
Statistical Analysis 2: Comparison: Positive Control Dentifrice (KNO3 Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); Test type: Superiority; p = 0.0761, Mixed Model with Repeated Measures; Least Square Mean Difference = -0.6447, 95% CI 2-sided [-1.3586 to 0.06924], Standard Error of Mean 0.3589 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Reference Dentifrice value
Statistical Analysis 3: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); Test type: Superiority; p = 0.9698, Mixed Model with Repeated Measures; Least Square Mean Difference = -0.01316, 95% CI 2-sided [-0.7031 to 0.6767], Standard Error of Mean 0.3469 — Least Square Mean Difference was calculated as Test Dentifrice value minus Reference Dentifrice value

12. Secondary Outcome: Mean Percentage of Tooth Sensitivity-free Days During Tooth Bleaching
Description: The tooth sensitivity questionnaire was used to describe the overall tooth sensitivity experienced by the participant during the previous 24 hours. Percentage of days during tooth bleaching where participants reported no tooth sensitivity in the tooth sensitivity questionnaire were reported.
Time Frame: Day 15 up to Day 21
Population: mITT population.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: percentage of days
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Number analyzed (Participants) | 31 | 27 | 30
percentage of days | 17.0 [12.2 to 23.8] | 19.0 [13.5 to 26.7] | 17.7 [12.7 to 24.8]

13. Secondary Outcome: Percentage of Days Analgesics Were Used to Alleviate Tooth Sensitivity During Tooth Bleaching
Description: The tooth sensitivity questionnaire was used to describe the overall tooth sensitivity experienced by the participant during the previous 24 hours. Percentage of days (derived for each participant) during tooth bleaching where participants reported the use of analgesics to relieve tooth sensitivity/pain in the tooth sensitivity questionnaire were reported.
Time Frame: Day 15 up to Day 21
Population: mITT population.
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Number analyzed (Participants) | 31 | 27 | 30
percentage of days | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

14. Secondary Outcome: Mean VAS Score Post Completion of Tooth Bleaching
Description: as for outcome 9
Time Frame: Day 22 up to Day 36
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: millimeter
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Number analyzed (Participants) | 31 | 27 | 30
millimeter | 25.0948 (4.0687) | 19.0720 (4.3244) | 28.4576 (4.0951)
Statistical Analysis 1: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Positive Control Dentifrice (KNO3 Containing Dentifrice); Test type: Superiority; p = 0.3142, Mixed Model with Repeated Measures; Least Square Mean Difference = -6.0228, 95% CI 2-sided [-17.8534 to 5.8078], Standard Error of Mean 5.9481 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Test Dentifrice value
Statistical Analysis 2: Comparison: Positive Control Dentifrice (KNO3 Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); Test type: Superiority; p = 0.1189, Mixed Model with Repeated Measures; Least Square Mean Difference = -9.3856, 95% CI 2-sided [-21.2335 to 2.4624], Standard Error of Mean 5.9568 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Reference Dentifrice value
Statistical Analysis 3: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); Test type: Superiority; p = 0.5612, Mixed Model with Repeated Measures; Least Square Mean Difference = -3.3627, 95% CI 2-sided [-14.8264 to 8.1009], Standard Error of Mean 5.7636 — Least Square Mean Difference was calculated as Test Dentifrice value minus Reference Dentifrice value

15. Secondary Outcome: Mean LMS Score Post Completion of Tooth Bleaching
Description: as for outcome 10
Time Frame: Day 22 up to Day 36
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: millimeter
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Number analyzed (Participants) | 31 | 27 | 30
millimeter
  LMS Intensity | 17.8845 (3.2466) | 16.9250 (3.4264) | 20.5072 (3.2181)
  LMS Duration | 17.4989 (2.6791) | 15.0944 (2.7983) | 19.2415 (2.6559)
  LMS Tolerability | 14.7900 (2.5500) | 15.4884 (2.7406) | 18.7096 (2.5932)
  LMS Description | 20.7559 (3.1888) | 18.2722 (3.4002) | 21.2502 (3.2253)
Statistical Analysis 1: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Positive Control Dentifrice (KNO3 Containing Dentifrice); LMS Intensity; Test type: Superiority; p = 0.8417, Mixed Model with Repeated Measures; Least Square Mean Difference = -0.9595, 95% CI 2-sided [-10.4856 to 8.5665], Standard Error of Mean 4.7895 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Test Dentifrice value
Statistical Analysis 2: Comparison: Positive Control Dentifrice (KNO3 Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); LMS Intensity; Test type: Superiority; p = 0.4487, Mixed Model with Repeated Measures; Least Square Mean Difference = -3.5821, 95% CI 2-sided [-12.9420 to 5.7777], Standard Error of Mean 4.7059 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Reference Dentifrice value
Statistical Analysis 3: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); LMS Intensity; Test type: Superiority; p = 0.5670, Mixed Model with Repeated Measures; Least Square Mean Difference = -2.6226, 95% CI 2-sided [-11.6970 to 6.4517], Standard Error of Mean 4.5624 — Least Square Mean Difference was calculated as Test Dentifrice value minus Reference Dentifrice value
Statistical Analysis 4: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Positive Control Dentifrice (KNO3 Containing Dentifrice); LMS Duration; Test type: Superiority; p = 0.5395, Mixed Model with Repeated Measures; Least Square Mean Difference = -2.4045, 95% CI 2-sided [-10.1672 to 5.3583], Standard Error of Mean 3.9029 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Test Dentifrice value
Statistical Analysis 5: Comparison: Positive Control Dentifrice (KNO3 Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); LMS Duration; Test type: Superiority; p = 0.2843, Mixed Model with Repeated Measures; Least Square Mean Difference = -4.1471, 95% CI 2-sided [-11.8005 to 3.5062], Standard Error of Mean 3.8479 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Reference Dentifrice value
Statistical Analysis 6: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); LMS Duration; Test type: Superiority; p = 0.6488, Mixed Model with Repeated Measures; Least Square Mean Difference = -1.7427, 95% CI 2-sided [-9.3255 to 5.8401], Standard Error of Mean 3.8124 — Least Square Mean Difference was calculated as Test Dentifrice value minus Reference Dentifrice value
Statistical Analysis 7: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Positive Control Dentifrice (KNO3 Containing Dentifrice); LMS Tolerability; Test type: Superiority; p = 0.8527, Mixed Model with Repeated Measures; Least Square Mean Difference = 0.6984, 95% CI 2-sided [-6.7589 to 8.1556], Standard Error of Mean 3.7493 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Test Dentifrice value
Statistical Analysis 8: Comparison: Positive Control Dentifrice (KNO3 Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); LMS Tolerability; Test type: Superiority; p = 0.3950, Mixed Model with Repeated Measures; Least Square Mean Difference = -3.2212, 95% CI 2-sided [-10.7149 to 4.2726], Standard Error of Mean 3.7677 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Reference Dentifrice value
Statistical Analysis 9: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); LMS Tolerability; Test type: Superiority; p = 0.2847, Mixed Model with Repeated Measures; Least Square Mean Difference = -3.9195, 95% CI 2-sided [-11.1588 to 3.3198], Standard Error of Mean 3.6397 — Least Square Mean Difference was calculated as Test Dentifrice value minus Reference Dentifrice value
Statistical Analysis 10: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Positive Control Dentifrice (KNO3 Containing Dentifrice); LMS Description; Test type: Superiority; p = 0.5954, Mixed Model with Repeated Measures; Least Square Mean Difference = -2.4837, 95% CI 2-sided [-11.7512 to 6.7839], Standard Error of Mean 4.6595 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Test Dentifrice value
Statistical Analysis 11: Comparison: Positive Control Dentifrice (KNO3 Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); LMS Description; Test type: Superiority; p = 0.5271, Mixed Model with Repeated Measures; Least Square Mean Difference = -2.9779, 95% CI 2-sided [-12.3044 to 6.3485], Standard Error of Mean 4.6891 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Reference Dentifrice value
Statistical Analysis 12: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); LMS Description; Test type: Superiority; p = 0.9138, Mixed Model with Repeated Measures; Least Square Mean Difference = -0.4942, 95% CI 2-sided [-9.5478 to 8.5593], Standard Error of Mean 4.5519 — Least Square Mean Difference was calculated as Test Dentifrice value minus Reference Dentifrice value

16. Secondary Outcome: Mean Bothersomeness NRS Score Post Completion of Tooth Bleaching
Description: as for outcome 11
Time Frame: Day 22 up to Day 36
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Number analyzed (Participants) | 31 | 27 | 30
score on a scale | 2.9902 (0.3059) | 2.7262 (0.3278) | 3.2306 (0.3114)
Statistical Analysis 1: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Positive Control Dentifrice (KNO3 Containing Dentifrice); Test type: Superiority; p = 0.5551, Mixed Model with Repeated Measures; Least Square Mean Difference = -0.2639, 95% CI 2-sided [-1.1500 to 0.6221], Standard Error of Mean 0.4455 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Test Dentifrice value
Statistical Analysis 2: Comparison: Positive Control Dentifrice (KNO3 Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); Test type: Superiority; p = 0.2714, Mixed Model with Repeated Measures; Least Square Mean Difference = -0.5044, 95% CI 2-sided [-1.4104 to 0.4016], Standard Error of Mean 0.4555 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Reference Dentifrice value
Statistical Analysis 3: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); Test type: Superiority; p = 0.5864, Mixed Model with Repeated Measures; Least Square Mean Difference = -0.2404, 95% CI 2-sided [-1.1160 to 0.6351], Standard Error of Mean 0.4402 — Least Square Mean Difference was calculated as Test Dentifrice value minus Reference Dentifrice value

17. Secondary Outcome: Mean Percentage of Tooth Sensitivity-free Days Post Completion of Tooth Bleaching
Description: The tooth sensitivity questionnaire was used to describe the overall tooth sensitivity experienced by the participant during the previous 24 hours. Percentage of days post completion of tooth bleaching where participants reported no tooth sensitivity in the tooth sensitivity questionnaire were reported.
Time Frame: Day 22 up to Day 36
Population: mITT population.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: percentage of days
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Number analyzed (Participants) | 31 | 27 | 30
percentage of days | 32.4 [19.2 to 54.7] | 41.3 [23.7 to 72.1] | 41.0 [24.3 to 69.1]

18. Secondary Outcome: Percentage of Days Analgesics Were Used to Alleviate Tooth Sensitivity Post Completion of Tooth Bleaching
Description: as for outcome 13
Time Frame: Day 22 up to Day 36
Population: mITT population.
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Number analyzed (Participants) | 31 | 27 | 30
percentage of days | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

19. Secondary Outcome: Change From Pre to Post-tooth Bleaching in Mean VITA Shade Score
Description: Tooth shade (color) of the facial surfaces of the anterior 6 maxillary and mandibular teeth were assessed by a single, trained clinical examiner using the VITA Bleachedguide 3D-MASTER. VITA Bleachedguide 3D-MASTER uses a value-ranked ordered scale from 1 (the lightest) to 29 (the darkest). The shade level of each tooth surface was scored visually by the clinical examiner with reference to the Bleachedguide. Lower scores indicated an improvement.
Time Frame: Day 15 (Pre-bleaching) up to Day 22 (Post-bleaching)
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
Number analyzed (Participants) | 31 | 27 | 30
score on a scale | -3.3043 (0.2877) | -3.6640 (0.3099) | -3.2813 (0.2927)
Statistical Analysis 1: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Positive Control Dentifrice (KNO3 Containing Dentifrice); Test type: Superiority; p = 0.3984, ANCOVA; Least Square Mean Difference = -0.3597, 95% CI 2-sided [-1.2026 to 0.4831], Standard Error of Mean 0.4238 — Least Square Mean Difference was calculated as Positive Control Dentifrice minus Test Dentifrice value
Statistical Analysis 2: Comparison: Positive Control Dentifrice (KNO3 Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); Test type: Superiority; p = 0.3734, ANCOVA; Least Square Mean Difference = -0.3827, 95% CI 2-sided [-1.2332 to 0.4678], Standard Error of Mean 0.4277 — Least Square Mean Difference was calculated as Positive Control Dentifrice value minus Reference Dentifrice
Statistical Analysis 3: Comparison: Test Dentifrice (NovaMin Containing Dentifrice) vs Reference Dentifrice (Regular Fluoride Dentifrice); Test type: Superiority; p = 0.9555, ANCOVA; Least Square Mean Difference = -0.02296, 95% CI 2-sided [-0.8382 to 0.7923], Standard Error of Mean 0.4099 — Least Square Mean Difference was calculated as Test Dentifrice value minus Reference Dentifrice value

ADVERSE EVENTS:
Time Frame: From signing of informed consent form until 5 days after last administration of study product or last study procedure (up to approximately 41 days).
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study product including any washout or lead-in product (or medical device), whether or not considered related to the study product, including any washout or lead-in product (or medical device). A serious AE (SAE) was a particular category of AE where the adverse outcome was serious.
Arm/Group | Test Dentifrice (NovaMin Containing Dentifrice) | Positive Control Dentifrice (KNO3 Containing Dentifrice) | Reference Dentifrice (Regular Fluoride Dentifrice)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 2/31 | 0/29 | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Dentifrice (NovaMin Containing Dentifrice) (N=31) | Positive Control Dentifrice (KNO3 Containing Dentifrice) (N=29) | Reference Dentifrice (Regular Fluoride Dentifrice) (N=30)
Headache (Nervous system disorders) | 1 | 0 | 2
Gingival Inflammation (Gastrointestinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT06608368/Prot_SAP_000.pdf